CLINICAL TRIAL: NCT00641628
Title: Subcutaneous Mastectomy With Conservation of the Nipple Areola Complex: Broadening the Indications
Brief Title: Nipple Areola Complex Conservation
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Stefan Paepke, MD, Technical University of Munich
Other Study IDs: NAC01
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
Keywords: Nipple sparing mastectomy; NAC conservation
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast Carcinoma Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: mastectomy

INTERVENTIONS:
Procedure: mastectomy
  Other Names: breast surgery

SUMMARY:
96 patients were offered a nipple sparing mastectomy.

DETAILED DESCRIPTION:
96 patients were operated on 109 breasts between Jul 2003 and May 2006 because of breast cancer, recurrence was observed.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer

Exclusion Criteria:

* inflammatory breast cancer
* clinical skin or nipple involvement

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
tumour recurrence | 07/2003 - 02/2008
% of nipple areola complex conservation | 07/2003 - 02/2008

SECONDARY OUTCOMES:
cosmetics
patient's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Marion Kiechle, MD, Study Chair — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Munich, Germany

REFERENCES:
- [Derived] Paepke S, Schmid R, Fleckner S, Paepke D, Niemeyer M, Schmalfeldt B, Jacobs VR, Kiechle M. Subcutaneous mastectomy with conservation of the nipple-areola skin: broadening the indications. Ann Surg. 2009 Aug;250(2):288-92. doi: 10.1097/SLA.0b013e3181b0c7d8. PMID 19638905